CLINICAL TRIAL: NCT01226888
Title: Prospective Study of Changes in Brown Adipose Tissue (BAT) Activity in Men Receiving Androgen Deprivation Therapy (ADT) With a GnRH Agonist or Antagonist for Prostate Cancer
Brief Title: Changes in Brown Adipose Tissue Activity In Men Receiving Androgen Deprivation Therapy for Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Philip J. Saylor, MD, Instructor, Massachusetts General Hospital
Other Study IDs: 10-037
Record Dates: First submitted 2010-10-04; First posted 2010-10-22 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Prostate Cancer
Keywords: brown adipose tissue; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fine needle aspirate biopsies of subcutaneous fat
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Androgen deprivation therapy (ADT) is considered standard of care for prostate cancer. However, changes in the patients metabolism are usually seen as a result of hormone therapy. These changes include increased fat mass, decreased lean mass, weight gain, high blood cholesterol, increased incidence of diabetes, and possibly increased incidence of cardiac events such as heart attack. The researchers of this trial would like to learn if these change in body mass are affected by the presence of brown fat in the body. Brown fat is made up of fat cells that are stored in the body and generate heat to control body temperature. Levels of brown fat are at the highest in newborn babies and decrease over time into adulthood. The researchers of this trial would like to learn more about these changes in metabolism during prostate cancer treatment by studying the changes in brown fat during the first 12 months of hormone therapy.

DETAILED DESCRIPTION:
* Participants will be asked to come into the clinic for additional visits before they begin hormone therapy. The following procedures will be performed: Cold-activated PET/CT scan; body composition DXA scan; blood tests, questionnaires and abdominal fat biopsy.
* During hormone therapy, the participant will return to the clinical once after 3 months, and again after 6 months, to draw blood for laboratory tests.
* After 12 months of hormone therapy, the participant will return to teh clinic to repeat the following procedures: Cold-activated PET/CT scan; body composition DXA scan; blood tests; questionnaires and abdominal fat biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Scheduled to initiate GnRH agonist or antagonist treatment with an intended treatment duration of 12 months or greater
* ECOG Performance status of 0 or 1
* Ability to understand and the willingness to sign a written informed consent
* 65 years of age or younger

Exclusion Criteria:

* Diagnosis of diabetes
* Ongoing corticosteroid use
* GnRH agonist or antagonist treatment within the last 2 years
* Ongoing beta-blocker use
* Body mass index of greater than 30

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men initiating androgen deprivation therapy with a GnRH agoinist or antagonist
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in brown adipose tissue activity | 1 year
  To assess the change in cold-activated borwn adipose tissue (BAT) activity upon initiation of GnRH agoinist or antagoinist therapy among men treated for prostate cancer. The primary endpoint is percent change in cold-activated BAT volumne after 12 months of treatment.

SECONDARY OUTCOMES:
Interval change | 1 year
  To describe interval change in total body weight and body mass during GnRH agonist or antagonist therapy.
Interval change | 1 year
  To describe interval change in Total body fat mass as determined by body composition dual energy x-ray absorptiometry (DXA) scan during GnRH agonist or antagonist therapy.
Interval change | 1 year
  To describe interval change in abdominal cross sectional subcutaneous fat area at the L4 verterbral body level during GnRH agonist or antagonist therapy.
Interval change | 1 year
  To describe interval change in insulin sensitivity (as refelcted by hemoglobin A1C, fasting plasma glucose, and fasting plasma insulin) during GnRH agonist or antagonist therapy.
Interval change | 1 year
  To describe interval change in serum lipid profile during GnRH agonist or antagonist therapy.
Interval change | 1 year
  To describe interval change in levels of several markers of BAT regulation & activity in abdominal subcutaneous fat during GnRH agonist or antagonist therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Saylor, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States